CLINICAL TRIAL: NCT00681408
Title: Omega 3 Fish Oil Supplements vs. Placebo for Patients With Non-alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Stephen Caldwell, MD, Professor, Department of Gastroenterology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12442; R21AT002901 (NIH); IRB # 12442; GCRC: SHC003; Grant # 5R21AT2901-2
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Non-alcoholic Steatohepatitis; Fatty Liver
Keywords: Steatohepatitis; NASH; NAFLD; omega 3 fatty acids; Exercise conditioning
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega 3 recipient arm (Active Comparator)
  Interventions: Drug: Omega 3 Fish Oil supplements
- Placebo (Placebo Comparator): Placebo fish oil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 Fish Oil supplements — Subjects in this arm will receive 3 grams daily Omega 3 fish oil supplements
  Other Names: Fish Oil capsules
  Arms: Omega 3 recipient arm
Drug: Placebo — Fish oil placebo pills
  Arms: Placebo

SUMMARY:
Nonalcoholic steatohepatitis (NASH) occurs in 2-3% of the US population and carries a 15-20% chance of progression to cirrhosis. It is closely associated with obesity, hyperlipidemia and insulin resistance. Therapy usually includes recommendations to increase exercise and to begin weight reducing diets but these goals are variably achieved and their relative effects in conjunction with pharmacological intervention have not been well defined. Moreover, these lifestyle changes can confound results of treatment trials if not quantified through conditioning testing and measures of body fat. Polyunsaturated fatty acids, especially formulation rich in omega-3, are widely accepted and endorsed in the medical community for their beneficial effects on hyperlipidemia and coronary disease risk reduction. Recent data suggests that omega-3 fatty acids ameliorate hepatic steatosis in humans and in animal models of NASH by reducing hepatic fat content. We hypothesize that a one year course of omega-3 fatty acid (3gm/day) will produce improvement in NASH histological injury independent of changes in weight (BMI) or degree of conditioning measured by the lactate threshold. The effects of the supplement will be compared to a placebo group and controlled for these lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

1. NASH with NAS (NASH Activity Score) of >4 evident on a biopsy performed within 6 months of enrollment.
2. Age 21 years or older.
3. BMI 25 or greater.
4. Ability to provide informed consent.

Exclusion Criteria:

1. Cirrhosis evident clinically or on biopsy.
2. Secondary forms of NASH such as that seen with bariatric surgery or medication induced from such medications as methotrexate, amiodarone, tamoxifen, corticosteroids.
3. Current or past history of diabetes or hyperlipidemia requiring specific drug therapy (see below).
4. Current use of a weight loss medicine, such as a 'fat-burner' or similar agent
5. Alcohol consumption > 30 g/day, currently or for more than 3 consecutive months within 5 years.
6. Other liver disease (hepatitis C,B, Wilson's, autoimmune, ct-1-antitrypsin and hemochromatosis or HIV
7. Pregnancy or unwillingness to use an effective form of birth control for women of child bearing years.
8. Renal insufficiency (creatinine > 2), symptomatic coronary, peripheral or neurovascular disease, symptomatic heart failure or advanced respiratory disease requiring oxygen therapy.
9. Inability to provide informed consent.
10. Any condition in the opinion of the primary investigator that would contraindicate the patient's participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The Primary endpoint will be improvement in a composite score of histological injury as measured by the NASH Activity Score (NAS). | approximately 12 months from enrollment

SECONDARY OUTCOMES:
Measurement of anthropometric indices (weight, BMI, waist circumference) | 12 months
Index of cardiorespiratory fitness determined by exercise tolerance (measured by lactate threshold on an exercise treadmill) | 12 months
Hepatic fat content measured by magnetic resonance imaging | 12 months
Changes in fasting plasma lipids, red cell fatty acid content, changes in anti-hyperlipidemia requirements, insulin sensitivity, and markers of inflammation including tumor necrosis factor and C-reactive protein | 12 mos

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Caldwell, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Argo CK, Patrie JT, Lackner C, Henry TD, de Lange EE, Weltman AL, Shah NL, Al-Osaimi AM, Pramoonjago P, Jayakumar S, Binder LP, Simmons-Egolf WD, Burks SG, Bao Y, Taylor AG, Rodriguez J, Caldwell SH. Effects of n-3 fish oil on metabolic and histological parameters in NASH: a double-blind, randomized, placebo-controlled trial. J Hepatol. 2015 Jan;62(1):190-7. doi: 10.1016/j.jhep.2014.08.036. Epub 2014 Sep 6. PMID 25195547